CLINICAL TRIAL: NCT04417881
Title: EVALUER L'IMPACT PREDICTIF DU SCORE MEESSI POUR LA STRATIFICATION DU RISQUE DES PATIENTS ADMIS POUR INSUFFISANCE CARDIAQUE AIGUE DANS LES STRUCTURES D'URGENCES (ICA-MEESSI)
Brief Title: EVALUER L'IMPACT PREDICTIF DU SCORE MEESSI POUR LA STRATIFICATION DU RISQUE DES PATIENTS ADMIS POUR INSUFFISANCE CARDIAQUE AIGUE DANS LES STRUCTURES D'URGENCES
Acronym: ICA-MEESSI
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7880
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Acurate Heart Failure
Keywords: caring; emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with acurate heart failure
  Interventions: Other: MEESSI score

INTERVENTIONS:
Other: MEESSI score — MEESSI score in predicting mortality and readmission of patients managed for acute heart failure (AHF) in Emergency Department.

SUMMARY:
Our primary purpose is to assess MEESSI score in predicting mortality and readmission of patients managed for acute heart failure (AHF) in Emergency Department.

European Society of Cardiology recommend risk stratification for patients with AHF. MEESSI score is not prospectively validated out of Spain.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient admitted to emergencies with suspicion of ICA according to the clinical intuition of the emergency doctor after interrogation, clinical examination, biology and imaging
* Patient with health insurance
* Subject who accept to participate in the research

Exclusion Criteria:

* Patient who refuse to participate in the study
* Patient with coronary syndrome with ST segment elevation
* Other diagnosis of dyspnea
* Persons deprived of their freedom or under the protection of justice
* Persons under guardianship or curatorship
* Impossibility of giving the patient informed information
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to emergencies with suspicion of ICA
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
MEESSI score | 30 days
  Tscore to predict the patient's future in the month following management for ED ICA. That is to say the number of days alive outside the hospital in the month following an ICA episode.

SECONDARY OUTCOMES:
Re-admission rate | 30 days
  30-day re-admission rate compared between the 4 risk categories defined by the MEESSI score
Mortality rate | 30 days
  Mortality rate at 30 days compared between the 4 risk categories defined by the MEESSI score
Sensitivity | 30 days
  Sensitivity, specificity and ROC curve of the MEESSI score in relation to the composite criterion according to the 4 risk categories

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Jean Rougié, Cahors
  - Hôpitaux Civils de Colmar, Colmar
  - CH Haguenau, Haguenau
  - Centre Hospitalier Forez, Montbrison
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU Pitié Salpetrière, Paris
  - CHU de Reims, Reims
  - CH Remiremont, Remiremont
  - Hôpital Robert Pax, Sarreguemines
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - Hôpital Nord Franche Comté, Trévenans

IPD SHARING:
Plan to Share IPD: Undecided